CLINICAL TRIAL: NCT05545696
Title: Comparison of Dental Arch Surface Scanning With and Without AI Support: A Methodological Study
Brief Title: Artificial Intelligence Supported Intraoral Scanning.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kıvanç Akça (Other)
Collaborators: Hacettepe University (Other)
Responsible Party: Sponsor-Investigator, Kıvanç Akça, Prof. Dr., Hacettepe University
Organization: Hacettepe University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: KA-21086
Record Dates: First submitted 2022-05-26; First posted 2022-09-19 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Impression Technic, Dental
Keywords: intraoral scanner; digitalization; Artificial intelligence

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI on scanning (Sham Comparator): The lower jaw of the participants was scanned with ''AI on'' scanning in line with recommended scanning protocol, and the IOS software automatically recorded the obtained data.
  Interventions: Device: AI on algorithm
- AI off scanning (Active Comparator): The lower jaw of the participants was scanned with ''AI off'' scanning in line with recommended scanning protocol, and the IOS software automatically recorded the obtained data.
  Interventions: Device: AI off algorithm

INTERVENTIONS:
Device: AI on algorithm — The mandibles of the participants were scanned with ''AI on'' scanning in line with the recommended scanning protocol. All scans were performed by the same operator.
  Arms: AI on scanning
Device: AI off algorithm — The mandibles of the participants were scanned with ''AI off'' scanning in line with the recommended scanning protocol. All scans were performed by the same operator.
  Arms: AI off scanning

SUMMARY:
Digitization (automation) of production stages with Computer-Aided Design and Computer-Aided Manufacturing (CAD/CAM) technologies has led to a digital revolution in dentistry, as in many other fields of the industry. In current dentistry, the digitalization process can be defined as direct and indirect workflow. The clinical reliability and success of the indirect digital workflow made possible by these technologies have been proven by scientific studies. With the development of intraoral scanners (IOS), a virtual model is obtained by direct digitalization. This method eliminated the conventıonale impression and dental cast model steps required for indirect digitalization. Intraoral scanners are used as an alternative to convantıonal impressions in single and short edentulous cases. It has already been emphasized that direct digitalization is a reliable alternative to the conventional impression method, as the clinical applicability, accuracy, and precision of the manufactured restorations have been scientifically verified. Therefore, the clinical use of direct digitalization is increasing (exponentially) day by day, and new upgraded versions of software, along with various modifications for the hardware equipment, are being developed. Integrating artificial intelligence (AI) supported software into the intraoral scanning process can be seen as the beginning of a new era for direct digitalization. Therefore the aim of this study is to evaluate the effect of artificial intelligence on the scanning time, the amount of data collected, and the image accuracy obtained.

DETAILED DESCRIPTION:
It was planned intraoral scanning (3Shape TRIOS A/S, Copenhagen, Denmark) of the participants' mandible (n=21) with artificial intelligence (AI on) and without artificial intelligence (AI off). Reference equilateral triangles for scanning were digitally designed and produced with a 3D printer. Then these triangles bonded to the buccal surfaces of #34, #44, and the lingual surfaces of #36#46 teeth. The lower jaw of each participant was scanned by the same operator, in line with the recommended scanning protocol. Furthermore, scanning was performed randomly, with AI on and off.

The IOS software automatically recorded the data required for quantitative comparing the scanning time and the obtained images (TRIOS Scanning Version 1.18.310, 3Shape A/S). In order to compare the scanning effectiveness between the methods, the area data of the digital images of the triangular objects obtained during both scans were calculated in a computer environment with reverse engineering software (Geomagic design X version 2016.1.0, 3D Systems Inc. Rock Hill, SC).

ELIGIBILITY:
Inclusion Criteria:

* Completed growth and development
* Good oral hygiene habits and healthy periodontal status.
* Absence of missing teeth in mandibula (or no teeth loss in mandibular)
* Signing of the informed consent form
* No temporomandibular joint (TMJ) disorder

Exclusion Criteria:

* Volunteers who are not fulfilling the inclusion criteria

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-10-10 (Actual); Study Completion 2021-12-05 (Actual)

PRIMARY OUTCOMES:
Scanning time and collected data | during the intraoral scanning
  The scanning time (in minutes and seconds) and the amount of collected data (as the count of images), automatically recorded by the intraoral scanning software, will be used to compare the two scanning methods.

SECONDARY OUTCOMES:
Surface area measurment of triangles | through study completion, an average of 2 weeks
  The area data of the triangular objects obtained during both scans were calculated in a computer environment with reverse engineering software.

CONTACTS AND LOCATIONS:
Overall Officials: Kivanc Akca, Professor, Study Director — Study Director
Locations (1):
- Hacettepe University Faculty of Dentistry Department of Prosthodontics, Ankara, Turkey (Türkiye)